CLINICAL TRIAL: NCT02611258
Title: Study on New Insights in Remodeling of Endocrine Cardiomyopathies: Intramyocardial, Molecular and Neuroendocrine Assessment in Response to Chronic Inhibition of Cyclic GMP Phosphodiesterase 5A in Cushing's Syndrome
Brief Title: Endocrine Cardiomyopathy in Cushing Syndrome: Response to Cyclic GMP PDE5 inhibitOrs
Acronym: ERGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrea M. Isidori (Other)
Responsible Party: Sponsor-Investigator, Andrea M. Isidori, MD - PhD, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERGO; 2015-004497-15 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Cushing's Syndrome Cardiomyopathy
Keywords: Left Ventricular Hypertrophy; Diastolic Dysfunction; Myocardial Fibrosis; Cushing's Syndrome
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Cushing Syndrome | interventions — Tadalafil

ARMS (1):
- Tadalafil (Experimental): Tadalafil 20 mg to be taken orally once daily, for 3 months
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Tadalafil 20 mg to be taken orally once daily, for 3 months
  Other Names: Cialis

SUMMARY:
Pathophysiology of Cushing's Syndrome (CS) cardiomyopathy is yet unclear and a specific treatment have not been indicated. It was already demonstrated the positive impact of phosphodiesterase type 5A (PDE5A) inhibition in several models of cardiomyopathy and in a model of endocrine cardiomyopathy due to type 2 diabetes mellitus. In this patients with diabetic cardiomyopathy it was demonstrated an improvement in cardiac kinetic, geometry and performance parameters and reduction of the ambulatory measurement of waist circumference.

This represents the first study that evaluate heart remodeling and performance changes and metabolic/immunological/molecular parameters after 5-months of Tadalafil 20 mg in Cushing's Syndrome cardiomyopathy. The proposed research will test whether phosphodiesterase 5A inhibition could become a new target for anti-remodeling drugs and to discover molecular pathways affected by this class of drugs and a network of circulating markers (miRNA) for the early diagnosis of Cushing's Syndrome cardiomyopathy.

The investigators hypothesize that:

* the signal molecules cGMP and cAMP could underlie the hypertrophic/profibrotic triggers related to this model of endocrine cardiomyopathy and that chronic inhibition of PDE5, activating cGMP signaling pathways, could improve cardiac remodeling due to CS;
* PDE5 inhibition could have a role in lipolytic regulation;
* neuroendocrine (e.g. natriuretic peptides) and metabolic markers and chemokines (e.g. MCP-1, TGF-ß) might relate with left ventricular remodeling in CS;
* there are neuroendocrine (e.g. natriuretic peptides), metabolic markers and chemokines (e.g. MCP-1, TGF-ß) related to cardiac disease in CS;
* miRNA expression [miR-208a, 499, 1, 133, 126, 29, 233, 222, 4454] might relate with left ventricular remodeling in CS;

DETAILED DESCRIPTION:
Mechanisms of action and evolutionary progression of Cushing's Syndrome (CS) cardiomyopathy are not yet been well elucidated and a specific treatment has not been identified. Our study aims to characterize the CS cardiomyopathy in terms of measuring the cardiac kinetic and performance parameters (tagged Cardiac Magnetic Resonance Imaging), fibrosis (T1-mapping technique). Our study will evaluate if PDE5A inhibition could become a new target for antiremodeling drugs in CS treated patients that developed cardiac hypertrophy and/or diastolic dysfunction independently of CS care accorded by current guidelines. The investigators also will explore the potential mechanisms of action of PDE5Ai: if exerted on cardiac tissue directly and contemporary also on other secondary pathways (analyzing vascular, endothelial, or metabolic markers).

A multidisciplinary approach will allow identifying a cluster of cardiovascular (NT-ProBNP, TGFb, MCP1) and metabolic indices, oxidative stress markers (iNOS, COX2, ROS, RANTES) and miRNAs, whose variations will analyze together with the CS cardiomyopathy parameters measured at CMR and 2D-echocardiography.

The Primary Objective is to evaluate the effects of PDE5Ai on Left Ventricular (LV) remodeling (kinetic and geometry parameters) at cine cardiac magnetic resonance (CMR) with tagging technique and contrast-enhanced and/or at 2D echocardiography with Tissue Doppler Imaging and speckle tracking in patients with CS cardiomyopathy

Secondary Objectives :

* to measure the effect of PDE5Ai on LV fibrosis at T1-mapping CMR at baseline and after PDE5Ai administration.
* to measure the effect of PDE5Ai on cardiac performance at cine CMR and at 2D echocardiography with Tissue Doppler Imaging and speckle tracking at baseline and after PDE5Ai administration.
* to measure the effect PDE5Ai of circulating cardiac-inflammatory-metabolic-endothelial molecular markers
* to measure the effect on bone and body composition

Patients will be screened at time 0. Follow up visits will take place every 4 weeks during treatment for 5 months and 1 month after the end of treatment.

Diagnostic procedures will include:

* physical examination with measurement of anthropometric parameters (weight, waist circumference, hip circumference) and vital signs (blood pressure, heart rate);
* blood sampling for assessing glucose and lipid metabolism, liver, renal, hematopoietic and coagulative function, thyroid and androgen hormones, ACTH and UFC, inflammatory parameters (cytokines, monocyte subpopulations) and microRNA;
* SF36, FSFI (in women), IEFF e IPSS (in men) questionnaires;
* cardiac exam, electrocardiogram and echocardiogram;
* MOC with DEXA;
* magnetic resonance imaging (MRI) with contrast-enhanced cardiac: T1-mapping for assessing cardiac fibrosis; tagging for evaluating kinetic parameters (torsion);

This is a pilot study proof-of-concept, then 10 patients are sufficient to detect the effect of PDE5Ai on cardiac remodeling in CS cardiomyopathy. Estimating a 80% drop-out of the study due to the complexity of CS and the related neuro-psychiatric involvement, 18 CS patients will be enrolled.

All variables will be tested for normality. Statistical analyzes will be performed using SPSS 18.0. The comparison before and after treatment will be made by non parametric Wilcoxon test. The investigators will calculate the confidence interval for the prevalence of the effect measured by χ2 test or Fisher exact test. The correlation was perfomed by Rho di Spearman.

ELIGIBILITY:
Inclusion Criteria:

* age>18 yrs;
* patients (men and women) with previous diagnosis of Cushing Syndrome (CS), surgically and/or clinically treated according to current guidelines, with stable parameters of CS disease in the last 3 months, and with concomitant cardiac hypertrophy and/or diastolic dysfunction developed independently of CS care and detected by 2D echocardiography;
* urinary free cortisol (UFC) levels in the normal range for sex and age;
* normal blood pressure or controlled hypertension

Exclusion Criteria:

* use of thiazolidinediones, or spironolactone; nitrates, doxazosin, terazosin e prazosin;
* current use of PDE5 inhibitors or previous (wash out of two months at least);
* congenital or valvular cardiomyopathy;
* recent ischemic heart disease or revascularization after a myocardial infarction (MI);
* contraindications to tadalafil use (hypersensitivity to tadalafil, nitrates use, severe cardiovascular disorders such as unstable angina or severe heart failure, severe hepatic impairment, blood pressure <90/50 mmHg, recent history of stroke or myocardial infarction and known hereditary degenerative retinal disorders such as retinitis pigmentosa);
* contraindications to CMR.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Change of Left ventricular torsion (°) | Baseline and 3 months after treatment
  Change of Left ventricular torsion (°) evaluated through Cardiac Magnetic Resonance

SECONDARY OUTCOMES:
Change of cardiac strain (σ - longitudinal shortening: strain %) | Baseline and 3 months after treatment
  Change of cardiac strain (σ - longitudinal shortening: strain %) evaluated through Cardiac Magnetic Resonance
Quantification of Myocardial fibrosis | Baseline and 3 months after treatment
  Quantification of Myocardial fibrosis assessed with T1-mapping through Cardiac Magnetic Resonance
Inflammatory indices | Baseline and 3 months after treatment
  Assessment of inflammatory indices (e.g. TGF-beta, MCP1)
Assessment of endothelial function markers Assessment of endothelial function markers | Baseline and 3 months after treatment
  Assessment of endothelial function markers (e.g ET-1, VEGF)
NT-proBNP | Baseline and 3 months after treatment
  Assessment of NT-proBNP
Assessment of oxidative stress markers | Baseline and 3 months after treatment
  Assessment of oxidative stress markers (eg iNOS, COX2, ROS, P Selectin, ICAM1)
cGMP | Baseline and 3 months after treatment
  Assessment of plasmatic levels of cGMP
Correlation analysis | Baseline and 3 months after treatment
  Correlation of biochemical parameters with cardiac parameters assessed through Cardiac Magnetic Resonance
Assessment of circulating microRNAs | Baseline
  Assessment of circulating microRNAs from plasma and white blood cells (miR208, 499, 1, 133, 29, 223, 222, 4454) and correlation of their levels to basal torsion, strain and fibrosis.
Changes of circulating miRNAs | Baseline and 3 months after treatment
  Changes of circulating miRNAs from plasma and white blood cells (miR208, 499, 1, 133, 29, 223, 222, 4454)
Assessment of circulating pro-fibrotic and pro-inflammatory chemokines | Baseline and 3 months after treatment
  Assessment of circulating pro-fibrotic and pro-inflammatory chemokines (MCP-1 and TGF-beta) and correlation to torsion, strain and fibrosis
Body composition | Baseline and 3 months after treatment
  Change of parameters of body composition evaluated by MOC with total body DEXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Giannetta, MD - Phd, Principal Investigator — Sapienza University of Rome, Policlinico Umberto I, Department of Experimental Medicine
Locations (1):
- Elisa Giannetta, Rome, Italy

REFERENCES:
- [Background] Giannetta E, Isidori AM, Galea N, Carbone I, Mandosi E, Vizza CD, Naro F, Morano S, Fedele F, Lenzi A. Chronic Inhibition of cGMP phosphodiesterase 5A improves diabetic cardiomyopathy: a randomized, controlled clinical trial using magnetic resonance imaging with myocardial tagging. Circulation. 2012 May 15;125(19):2323-33. doi: 10.1161/CIRCULATIONAHA.111.063412. Epub 2012 Apr 11. PMID 22496161
- [Background] Bernardo BC, Weeks KL, Pretorius L, McMullen JR. Molecular distinction between physiological and pathological cardiac hypertrophy: experimental findings and therapeutic strategies. Pharmacol Ther. 2010 Oct;128(1):191-227. doi: 10.1016/j.pharmthera.2010.04.005. Epub 2010 May 12. PMID 20438756
- [Background] Montgomery RL, Hullinger TG, Semus HM, Dickinson BA, Seto AG, Lynch JM, Stack C, Latimer PA, Olson EN, van Rooij E. Therapeutic inhibition of miR-208a improves cardiac function and survival during heart failure. Circulation. 2011 Oct 4;124(14):1537-47. doi: 10.1161/CIRCULATIONAHA.111.030932. Epub 2011 Sep 6. PMID 21900086
- [Background] Fichtlscherer S, Zeiher AM, Dimmeler S. Circulating microRNAs: biomarkers or mediators of cardiovascular diseases? Arterioscler Thromb Vasc Biol. 2011 Nov;31(11):2383-90. doi: 10.1161/ATVBAHA.111.226696. PMID 22011751
- [Background] Baseler WA, Thapa D, Jagannathan R, Dabkowski ER, Croston TL, Hollander JM. miR-141 as a regulator of the mitochondrial phosphate carrier (Slc25a3) in the type 1 diabetic heart. Am J Physiol Cell Physiol. 2012 Dec 15;303(12):C1244-51. doi: 10.1152/ajpcell.00137.2012. Epub 2012 Oct 3. PMID 23034391
- [Background] De Leo M, Pivonello R, Auriemma RS, Cozzolino A, Vitale P, Simeoli C, De Martino MC, Lombardi G, Colao A. Cardiovascular disease in Cushing's syndrome: heart versus vasculature. Neuroendocrinology. 2010;92 Suppl 1:50-4. doi: 10.1159/000318566. Epub 2010 Sep 10. PMID 20829618